CLINICAL TRIAL: NCT03990974
Title: Postoperative Antimicrobial Prophylaxis Versus Placebo for Infection Prevention in Hepatocellular Carcinoma After Liver Resection: A Multi-center, Randomized, Open-labelled Trial.
Brief Title: Postoperative Antimicrobial Prophylaxis Versus Placebo for Infection Prevention in HCC After Liver Resection
Acronym: HCC
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: There were difficulties in implementation
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Kuang, Professor, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 20190236
Record Dates: First submitted 2019-06-18; First posted 2019-06-19 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Hepatocellular Carcinoma; Postoperative Infection
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Postoperative antimicrobial prophylaxis (Experimental): Patients will receive postoperative antimicrobial prophylaxis for 3 days in 24 hours after hepatectomy.
  Interventions: Drug: postoperative antimicrobial prophylaxis
- No postoperative antimicrobial prophylaxis (Sham Comparator): Patients will receive no antibiotics after hepatectomy, unless the clinicians suggest he/she need antibiotics to treat or prevent infection.
  Interventions: Other: No postoperative antimicrobial prophylaxis

INTERVENTIONS:
Drug: postoperative antimicrobial prophylaxis — The drugs are all common antibiotics used to prevent postoperative infection in each hospital.
  Arms: Postoperative antimicrobial prophylaxis
Other: No postoperative antimicrobial prophylaxis — Patients will receive no antibiotics after hepatectomy unless necessary.
  Arms: No postoperative antimicrobial prophylaxis

SUMMARY:
This trial is a multi-center, double-blinded, randomized (1:1) clinical trial. The aim is to compare the postoperative infection rate between the 3 days postoperative AMP group and the placebo group in HCC patients undergoing hepatectomy.

DETAILED DESCRIPTION:
This trial includes two phase. The first phase is the internal pilot study to explore the expulsion rate and recruited population. The second phase is the main phase III trial.

ELIGIBILITY:
Inclusion Criteria:

* Age: over 18 years;
* Diagnosed as primary HCC according to the EASL criteria and plan to receive hepatectomy;
* Child-Pugh A class;
* No history of antibiotics in 1 week before surgery, except for antimicrobial prophylaxis in the 24h before surgery.
* No evidence of infection during preoperational assessment

Exclusion Criteria:

* Underwent hepatectomy combined with resection of other organs, except for gallbladder;
* Found obvious infection during operation;
* Combination with other operations, such as biliary reconstruction or tube drainage, bile duct exploration and stone remove, etc.;
* Allergic to the antibiotics used in the 24h before surgery;
* Emergency surgery;
* Tumor rupture;
* Did not underwent hepatectomy because of any reasons;
* Admission to ICU after surgery;
* ASA grade ≥ 3;
* Denial of informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
30-day postoperative infection rate | 30 days after hepatectomy
  the incidence rate of postoperative infection occurred in 30 days after surgery, including surgical site infections, distant infection or infection from unknown sources

SECONDARY OUTCOMES:
Surgical site infection rate | 30 days after hepatectomy
  the incidence rate of surgical site infection, including infections of the incision or organ or space that occur after surgery.
Postoperative complication rate | 3 months after hepatectomy
  the incidence rate of postoperative complications, grading as Clavien-Dindo grades
Severe infection rate | 30 days after hepatectomy
  the incidence rate of postoperative complications over grade 3
Distant infection rate | 30 days after hepatectomy
  the incidence rate of distant infections, including respiratory system infection, urinary system infection, catheter related infections or sepsis (defined as fever (temperature ≥38 ℃) or elevated white blood cell (> 10 x10^9 / L) accompanied by sputum, urine, catheter secretions, or blood culture positive.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China